CLINICAL TRIAL: NCT02620423
Title: A Phase 1b Study of Pembrolizumab (KEYTRUDA®) in Combination With REOLYSIN® (Pelareorep) and Chemotherapy in Patients With Advanced Pancreatic Adenocarcinoma
Brief Title: Study of Pembrolizumab With REOLYSIN® and Chemotherapy in Patients With Advanced Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REO 024
Record Dates: First submitted 2015-11-25; First posted 2015-12-03 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic; Cancer; REOLYSIN®; Chemotherapy; Pembrolizumab; KEYTRUDA®; Pelareorep; Reovirus; Oncolytic virus
MeSH Terms: conditions — Neoplasms | interventions — reolysin; Drug Therapy; Gemcitabine; Irinotecan; Leucovorin; Fluorouracil; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: REOLYSIN® — 4.5x10E10 TCID50 1 hour intravenous infusion, administered on Day 1 and 2 of a 21-day cycle
  Other Names: Pelareorep
Drug: Chemotherapy — Patients may be treated with one of three chemotherapy backbone regimens. The decision on the chemotherapy backbone is based on physician preference.This includes either: a) Gemcitabine or b) Irinotecan or c)Leucovorin followed by 5-fluorouracil
Drug: Gemcitabine — 1000 mg/m2 intravenous infusion over 30 minutes on Day 1 of a 21-day cycle or
Drug: Irinotecan — 125 mg/m2 intravenous infusion over 90 minutes on Day 1 of a 21-day cyle or
Drug: Leucovorin — Leucovorin (LV) followed by 5-fluorouracil (5FU). LV 200 mg/m2 intravenous infusion over 2 hours on Day 1, 5FU 200 mg/m2 intravenous infusion bolus over 5-10 minutes on Day 1, followed by 5FU 1200 mg/m2 continuous intravenous infusion over 22 hours on Day 1 of a 21-day cycle
Drug: 5-fluorouracil — Leucovorin (LV) followed by 5-fluorouracil (5FU). LV 200 mg/m2 intravenous infusion over 2 hours on Day 1, 5FU 200 mg/m2 intravenous infusion bolus over 5-10 minutes on Day 1, followed by 5FU 1200 mg/m2 continuous intravenous infusion over 22 hours on Day 1 of a 21-day cycle
Drug: Pembrolizumab — Pembrolizumab, 2 mg/kg intravenous infusion 30 minutes on Day 8 of a 21-day cycle
  Other Names: KEYTRUDA®

SUMMARY:
The purpose of this Phase 1b study is to investigate whether intravenous administration of REOLYSIN® in combination with chemotherapy and pembrolizumab is effective and safe in the treatment of pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Reovirus Serotype 3 - Dearing Strain (REOLYSIN®) is a naturally occurring, ubiquitous, non-enveloped human reovirus. It's primary mode of activity is to infect and selectively target tumors with activating Ras pathway mutations. Up to 70% of pancreatic cancers have activating Ras pathway mutations and/ or over-expressions.

This is an open label, Phase 1b study of REOLYSIN® and chemotherapy in combination with pembrolizumab in patients with advanced (unresectable or metastatic) histologically confirmed pancreatic adenocarcinoma that progressed after (or did not tolerate) first-line therapy. It is thought that Reovirus when combined with chemotherapy would lead to increased viral replication and oncolysis preferentially in RAS activated tumors, with resulting immunogenic response than can be further enhanced by checkpoint inhibition using pembrolizumab. The study is designed to characterize the efficacy and safety of REOLYSIN® given intravenously in combination with one of the three chemotherapy backbone regimens, Gemcitabine, Irinotecan or Leucovorin/ 5-fluorouracil (5-FU), and pembrolizumab, the treatment cycle of which will be repeated every 3 weeks. It will follow a 3+3 design with no dose escalations. 3 patients will be initially enrolled. If no dose limiting toxicities (DLT) are observed, the cohort will be expanded. Provided patients do not develop intolerable toxicity (that does not respond to either supportive care or dose reduction) or clinically meaningful disease progression, treatment with additional cycles may be continued so long as patients experience clinical benefit in the judgement of the Investigator.

ELIGIBILITY:
Inclusion Criteria: Each patient MUST:

* Have histologically confirmed advanced or metastatic pancreatic adenocarcinoma and have failed or did not tolerate first-line therapy.
* Have either archival tissue available for immune testing OR if not, a baseline biopsy of a primary or metastatic lesion (including ascites) which is accessible for a biopsy that can be accomplished with reasonable safety.
* Be available and agree to; a post-treatment tumor biopsy of either a primary or metastatic lesion (including ascites).
* Have measurable disease.
* Have no continuing acute toxic effects (except alopecia) of any prior anticancer treatment, i.e., all such effects must have resolved to Common Terminology Criteria for Adverse Events (CTCAE), version 4.02 [2], Grade ≤1. Any major surgery (except biopsies) must have occurred at least 28 days prior to study enrolment.
* Have an ECOG Performance Score ≤ 2.
* Have baseline laboratory results as follows:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10E9 [SI units 10E9/L].
  * Platelets ≥ 100 x10E9 [SI units 10E9/L] (without platelet transfusion)
  * Serum creatinine ≤ 1.5 x ULN.
  * Creatinine clearance (measured over 24 hours) OR calculated creatinine clearance (Cockcroft-Gault formula) of ≥ 60 mL/min.
  * Bilirubin ≤ 1.5 x ULN.
  * AST/ALT ≤ 3 x ULN (≤ 5 x ULN if patients have liver metastasis).
  * TSH, T4 and ACTH must be within normal range.
  * Proteinuria with normal or grade 1 OR Urinary protein < 1 g/24hr.
  * Negative pregnancy test for females of childbearing potential.
* Have signed an informed consent indicating that the patient is aware of the neoplastic nature of their disease and have been informed of the procedures of the protocol, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
* Be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests.

Exclusion Criteria: Each patient MUST NOT:

* Receive concurrent therapy with any other investigational anticancer agent while on study.
* Be on immunosuppressive therapy or have known HIV infection or active hepatitis B or C.
* Receive radiotherapy within 28 days prior to receiving study drug.
* Be a pregnant or breast-feeding woman. Female patients of childbearing potential must agree to use effective contraception, must be surgically sterile, or must be postmenopausal. Male patients must agree to use effective contraception or be surgically sterile. Barrier methods are a recommended form of contraception.
* Have clinically significant cardiac disease (New York Heart Association, Class III or IV) including pre-existing arrhythmia, uncontrolled angina pectoris, myocardial infarction 1 year prior to study entry, or grade 2 or higher compromised left ventricular ejection fraction.
* Have dementia or altered mental status that would prohibit informed consent.
* Have any other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal Investigator, would make the patient inappropriate for this study.
* Have HIGH BURDEN/SYMPTOMATIC brain metastases. LOW VOLUME / ASYMPTOMATIC and pre-treated clinically stable brain metastases ARE allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12; Primary Completion 2018-03 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Determine the safety and DLTs of REOLYSIN® and chemotherapy (gemcitabine OR irinotecan OR 5FU) in combination with pembrolizumab in patients with advanced pancreatic adenocarcinoma who have progressed after (or did not tolerate) first line treatment | During the first cycle of treatment (3 week cycle)

SECONDARY OUTCOMES:
Determine the overall response rate (ORR), and progression-free survival (PFS) by immune-related response criteria, as well as overall survival (OS) | Assessed every 9 weeks until disease progression or death. Post treatment scans every 3 months, if applicable.
Determine the effects of REOLYSIN® and pembrolizumab when administered in combination as determined by analysis of pre- and post-treatment biopsies and blood based immune markers | Biopsies (or available archival tumor tissue) performed before treatment begins and post treatment between Cycle 2 Day 15 and Cycle 3 Day 1. Immune marker analysis performed at start of treatment, Cycle 1 Day 1, Cycle 1 Day 8 and Cycle 2 Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sukeshi Patel Arora, MD, Principal Investigator — Cancer Therapy & Research Center at UTHSCSA
Locations (1):
- Cancer Therapy & Research Center at UTHSCSA, San Antonio, Texas, United States